CLINICAL TRIAL: NCT05853861
Title: Promoting Early Intervention Timing and Attention to Language
Acronym: PETAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor/PhD, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-001637
Record Dates: First submitted 2023-04-25; First posted 2023-05-11 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: MONITOR; COACH
Keywords: autism; siblings; JASPER; speech; intervention
MeSH Terms: conditions — Autistic Disorder; Speech | interventions — Activator Appliances

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MONITOR (No Intervention): Participants in this arm will be provided with information to track the early development of their infants, along with specific developmentally targeted activities.
- COACH (Experimental): Participants will be provided with a blended intervention of two evidence tested intervention, JASPER and Babble Bootcamp along with continued monitoring.
  Interventions: Behavioral: JASPER; Behavioral: Babble Bootcamp

INTERVENTIONS:
Behavioral: JASPER — JASPER is an evidence based early intervention that focuses on the core social communication and engagement skills of young children that are important to improvements in communication and language.
  Arms: COACH
Behavioral: Babble Bootcamp — Babble Bootcamp is a new intervention focusing on the speech-motor system and aims to improve babbling and early word use in infants known to be at risk for language delay.
  Arms: COACH

SUMMARY:
The proposed study (PETAL: Promoting Early intervention Timing and Attention to Language) aims to determine the timing of intervention among infants with Increased Likelihood for Autism (ILA; at risk for autism by virtue of having an older sibling with autism) on communication and language outcomes at 24 months. Results of this study will determine when (9 vs 12 vs 15 months), and based on which measures (brain, language, or their combination) to augment parental support with a specialized parent-mediated coaching intervention for optimal outcomes on communication and language at 24 months.

Children will be recruited at 6-8 months of age and will begin with entry assessments. All children will first begin with the MONITOR condition (using Ages & Stages Questionnaire (ASQ-3) and activity cards. Then when the child is 9 months, they will be randomized to continue with MONITOR condition or COACH condition (incorporates JASPER intervention and Babble Bootcamp) after second set of assessments. There are a total of 6 assessment timepoints (6-8 months of age, 9 months of age, 12 months of age, 15 months of age, 18 months of age, and 24 months of age). At time points of 9months and 12 months, the child will be randomized to COACH or MONITOR conditions. Once the child is randomized to COACH condition, they will continue with that condition until they terminate the study at 24 months. At the 15 months timepoint, there will no longer be a randomization. Children that were in the MONITOR condition will change to the COACH condition until they terminate the study.

DETAILED DESCRIPTION:
A total of 140 infants aged 6-8 months old who are siblings of children with ASD will participate, with an expected 30-60infants recruited each year for 3 years. We expect to recruit a diverse sample of ILA infants and families in two sites, LosAngeles area and Boston area; many will be from traditionally marginalized and minoritized families, mostly low income.Referrals will be elicited from community partners with which both sites have a long history, including school systems,federally qualified health centers, local clinics, family resource centers, and family support groups.

This study will use a four phase, Sequential Multiple Assignment Randomized Trial (SMART) design to examine theeffectiveness of transitioning to more intensive early intervention prior to 15 months of age, and to inform clinical decision-making concerning the optimal time to transition to more intensive intervention based on the specific characteristics of thechild. Phase 1 begins at age 6 months; after baseline demographic, language, behavior and brain assessments, allchildren are offered the MONITOR intervention. Phase 2 begins at age 9 months; after language, behavior and brainassessments, all children are randomly assigned to transition to MONITOR plus COACH (with probability 1/3) versuscontinue with MONITOR (with probability 2/3). Phase 3 begins at age 12 months; following language, behavior, and brainassessments, children who have not yet transitioned to MONITOR plus COACH are randomly assigned (with equalprobability) to transition to MONITOR plus COACH versus continue with MONITOR. Phase 4 begins at age 15 months;following language and behavior assessments, all remaining children will transition to MONITOR plus COACH.

The MONITOR condition consists will take a global, general domain approach to providing parents with information totrack the early development of their infants, along with specific developmentally targeted activities. The well validatedAges and Stages-3+ screening tool along with activity cards will provide information to parents at each age. All parentswill receive these materials at 3-month intervals, along with a developmentally chosen toy and book for their infant. Wewill provide an appropriate toy/book given we expect a diverse sample including many low resourced families. Thequestionnaire takes 10- 15 minutes to complete and covers developmental domains of communication, motor, problem-solving and personal-social, and is available in English, Spanish, and several other languages. We will drop off or mail thespecific form and activity card (plus toy and book) to families at each of our specified ages---6, 9, 12, 15, 18, 21 and 24months. The intervention activities card includes suggestions for games and other fun events for parent- infant dyads.Moreover, each family will have access to the intervention team (text, call, zoom) on an as needed protocol, and we willkeep track of all contact. The MONITOR intervention continues for all infants and parents throughout the study periodeven after receiving COACH intervention.

The COACH condition consists of a blended intervention of two evidence tested interventions, JASPER and BabbleBootcamp Infant-parent dyads will be randomized to receive COACH (JASPER Babble) at 9, 12 or 15 months. JASPERBabble addresses early parent-child social communication by helping to close the 'feedback loop'. When parents talk andplay with their infant, the infant increases their developmental behaviors which serve to provide more opportunities forparents to respond. Babble Bootcamp targets on babbling specifically will be incorporated into this feedback loop, and theimportance of the blended intervention should be underscored, providing both context and targets. For infant-parentdyads randomized to COACH, we will set up once weekly remote (zoom) 1-hour coaching sessions in betweenassessment visits each 3 months. Similar to the ASQ-3+ monitoring intervention, parents will have access to theintervention team on as needed basis throughout the study if they request more input, and we will track this contact. Oncerandomized to COACH, parents will continue to receive the remotely delivered intervention throughout the study period.

Assessments will be administered at 6 timepoints. At entry (when child is 6-8 months), parents will sign consent, fill outdemographic forms, treatment history form, Mullen, PCX, LENA, and EEG.

At the 9 months and 12 months timepoints, the Mullen, PCX, LENA, and EEG will be administered again.

At 15, 18, and 24 months, the Mullen, PCX, LENA will be administered. An ADOS-2 will also be administered at 24months only.

ELIGIBILITY:
Inclusion Criteria:

* This study will recruit approximately 140 infants ages 6-8 months of age who are younger siblings of children with ASD.
* Both males and females are eligible for study participation and will be recruited.
* Family income is under the very low income described under the Department of Housing and Community DevelopmentDivision of Housing Policy Agreement for the city of Los Angeles.

Exclusion Criteria:

* Infants who have seizures and are not stable on anti-seizure medication
* Infant is expected to have surgery over the next year
* Infant has associated physical disorders, and/or co-morbid with other syndromes or diseases.
* All of the children will be free of additional sensory or motor impairments (e.g., Visual or hearing impairment) and othergenetic syndromes (e.g., Down Syndrome).
* In addition, infants who are premature or less than 34 weeks (gestational age <34 weeks) will be excluded.

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Mullen Early Learning Scales (MSEL) | child's 6,9,12,15,18 and 24 months of age
  The MSEL provides expressive language scale T-scores. We will compare the changes in T-scores throughout the different time points, expecting improvement throughout each time point.

SECONDARY OUTCOMES:
Parent-Child Interaction (PCX) | child's 6,9,12,15,18 and 24 months of age
  A 15-minute parent-child play-based interaction will be collected at every time point. Expressive language (canonical babble ratio, number of different consonants, vocalizations and number of words), communicative gestures, joint engagement, and object play will be measured and compared at each time point.
LENA | child's 6,9,12,15,18 and 24 months of age
  Parents will collect day-long naturalistic recordings of their child's language environment. We will compare them throughout each time point.
Resting electroencephalogram test (EEG) | child's 6,9,12 months of age
  EEG data (L Fronto-Temporal (alpha, gamma)- coherence) will be recorded in the participants' home. They will be compared at the distinct time frames they are collected.

OTHER OUTCOMES:
Autism Diagnostic Observation Schedule-2 (ADOS-2) | 24 months of age
  At 24 months the ADOS (Mod 1 and 2) will be administered to determine diagnosis of autism.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - University of Massachusetts Medical Center, Worcester, Massachusetts

DOCUMENTS (1):
  • Informed Consent Form (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT05853861/ICF_000.pdf